CLINICAL TRIAL: NCT00941044
Title: Unloading of the Respiratory Muscles Using Non-invasive Neurally Adjusted Ventilatory Assist in Healthy, Resistively Loaded Volunteers
Brief Title: Non-invasive Neurally Adjusted Ventilatory Assist in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Lukas Brander, MD, University Hospital - Inselspital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KEK BE 062/09
Record Dates: First submitted 2009-07-16; First posted 2009-07-17 (Estimated); Last update posted 2010-02-05 (Estimated); Status verified 2010-02

CONDITIONS: Healthy
Keywords: non-invasive ventilation; diaphragm; electrical activity; neurally adjusted ventilatory assist; volunteers
MeSH Terms: interventions — Interactive Ventilatory Support

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- non-invasive NAVA (Experimental): application of non-invasive neurally adjusted ventilatory assist in healthy volunteers
  Interventions: Device: Neurally adjusted ventilatory assist

INTERVENTIONS:
Device: Neurally adjusted ventilatory assist — application of non-invasive NAVA in healthy volunteers

SUMMARY:
Neurally adjusted ventilatory assist (NAVA) is a new concept of mechanical ventilation. NAVA delivers assistance to spontaneous breathing based on the detection of the electrical activity of the diaphragm. The investigators will study the effects of non-invasive NAVA in respiratory muscle unloading in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Subject has given written informed consent.
* Male or female, aged 18 - 80 years (extremes included).

Exclusion Criteria:

* Pregnant or breast-feeding female. A pregnancy test will be performed in all female volunteers less than 60 yrs of age.
* Known intolerance or allergy against local anesthetic drugs such as procain, lidoocaine, xylocain.
* Any contraindication to the insertion of a nasogastric tube, including (but not limited to): severe oropharyngeal malformation or bleeding; esophageal varices, tumor, infection, stenosis, or rupture, bleeding disorder with evidence of active bleeding.
* Presence or suspicion of diaphragm injury.
* Prior medical history that might contribute to a disturbance of the neural system, including, but not limited to: diabetes, prior critical illness, carcinoma, uremia, vitamin B12 deficiency, chronic liver disease, alcohol abuse, malabsorption (sprue), HIV, Lyme disease, Lymphoma, multiple myeloma, hypothyroidism, systemic vasculitis, abnormalities on physical examination of peripheral nervous system (pallesthesia, impaired muscle strength according to the MRC Scale for Muscle Examination in 12 Muscle groups).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
changes in mean inspiratory airway pressure | beginning to end of study

SECONDARY OUTCOMES:
changes in respiratory pattern | begin to end of study

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Intensive Care Medicine, University Hospital - Inselspital, Bern, Canton of Bern, Switzerland

REFERENCES:
- [Background] Sinderby C, Navalesi P, Beck J, Skrobik Y, Comtois N, Friberg S, Gottfried SB, Lindstrom L. Neural control of mechanical ventilation in respiratory failure. Nat Med. 1999 Dec;5(12):1433-6. doi: 10.1038/71012. No abstract available. PMID 10581089
- [Derived] Tuchscherer D, Z'graggen WJ, Passath C, Takala J, Sinderby C, Brander L. Neurally adjusted ventilatory assist in patients with critical illness-associated polyneuromyopathy. Intensive Care Med. 2011 Dec;37(12):1951-61. doi: 10.1007/s00134-011-2376-0. Epub 2011 Nov 3. PMID 22048718